CLINICAL TRIAL: NCT03685630
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Tolerability of Intravenous Brivaracetam as Replacement for Oral Brivaracetam in Japanese Subjects >=16 Years of Age With Partial Seizures With or Without Secondary Generalization
Brief Title: A Study to Evaluate the Safety and Tolerability of Intravenous Brivaracetam (BRV) as Replacement for Oral Brivaracetam in Japanese Subjects >=16 Years of Age With Partial Seizures With or Without Secondary Generalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0118
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Partial Seizures With or Without Secondary Generalization; Epilepsy
Keywords: Brivaracetam; Epilepsy; Partial seizures with or without secondary generalization; Japanese subjects
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brivaracetam (Experimental): Subjects in this arm will receive open-label Brivaracetam.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — * Pharmaceutical form: Solution for injection
  * Concentration: 10 mg/ml
  * Route of administration: Intravenous injection
  Other Names: Briviact

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of intravenous (iv) brivaracetam (BRV) as adjunctive therapy administered as a replacement for oral BRV at doses ranging from BRV 50 mg/day to 200 mg/day in Japanese subjects >=16 years of age with partial seizures with or without secondary generalization and to evaluate the partial seizure frequency after switching from oral administration to iv BRV.

ELIGIBILITY:
Inclusion Criteria:

* Subject has, in the opinion of the Investigator, adequate seizure control for participation in the study, and is willing and able to comply with all study requirements including hospitalization, multiple blood draws, and intravenous (iv) injection
* Female subjects without childbearing potential (postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible. Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method
* Japanese subject is currently enrolled in EP0085 [NCT03250377] receiving oral brivaracetam (BRV) for the treatment of partial seizures and has been enrolled for at least 8 weeks prior to entry into EP0118
* Subject has been on a stable twice daily dosage regimen of BRV 50 mg/day to 200 mg/day for the 4 weeks prior to entry into EP0118
* Subject has been receiving concomitant antiepileptic drug (AED(s)) at doses that have remained stable for the 4 weeks (12 weeks for phenobarbital, phenytoin, and primidone) prior to entry into EP0118
* Subject has been receiving drugs with possible central nervous system (CNS) effects at doses that have remained stable for the 4 weeks prior to entry into EP0118, if applicable
* Subject has been receiving drugs that significantly influence the metabolism of BRV at doses that have remained stable for the 4 weeks prior to entry into EP0118, if applicable
* Subject has had stable vagal nerve stimulation (VNS) settings for the 4 weeks prior to entry into EP0118, if applicable

Exclusion Criteria:

* Subject is receiving an investigational medicinal product (IMP) or unapproved medication other than oral BRV, or using an experimental medical device
* Subject has previously been treated with intravenous (iv) brivaracetam (BRV)
* Subject has a known hypersensitivity to any components of the investigational medicinal product (IMP) or comparative drugs as stated in this protocol
* Subject has a confirmed clinically relevant abnormality by electrocardiogram (ECG)
* Subject has a severe medical, neurological, or psychiatric disorder, or abnormal laboratory values which may have an impact on the safety of the subject
* Subject has demonstrated poor compliance with the visit schedule or medication intake in previous BRV studies
* Subject has planned participation in any other clinical study of another IMP or device during this study
* Subject is a pregnant or lactating female
* Subject has any medical condition which, in the Investigator's opinion, warrants exclusion
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) "Since Last Visit" at Screening
* Subject has >2x upper limit of normal (ULN) of any of the following prior to Day 1 (from liver function assessment in EP0085): alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (>=1.5x ULN total bilirubin if known Gilbert's syndrome)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) as reported spontaneously by the subject or observed by the Investigator | From study entry until Final Visit (up to 7 days)
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Subject withdrawal due to Adverse Events (AEs) | From study entry until Final Visit (up to 7 days)
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Occurrence of Serious Adverse Events (SAEs) | From study entry until Final Visit (up to 7 days)
  A SAE must meet 1 or more of the following criteria:
  * Death
  * Life-threatening
  * Significant or persistent disability/incapacity
  * Congenital anomaly/birth defect
  * Initial inpatient hospitalization or prolongation of hospitalization
  * Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious

SECONDARY OUTCOMES:
Partial seizure frequency during the Treatment Period | During the Treatment Period (from Day 1 to Day 5)
  Partial Seizures can be classified into one of the following three groups: Simple Partial Seizures, Complex Partial Seizures, Partial Seizures evolving to Secondarily Generalized Seizures. The partial seizure frequency will be assessed using the seizure count information recorded on the daily record card (DRC). The written information will be discussed with the subject in order to ensure completeness and accuracy. As a result of the discussion, the Investigator will assess the seizures according to the International League Against Epilepsy (ILAE) codes and record the seizure types and frequency on the DRC.
Brivaracetam (BRV) plasma concentration (at Day 1) | Day 1
  The plasma concentration level of brivaracetam 5 minutes postdose on Day 1.
Brivaracetam (BRV) plasma concentration (at Day 2) | Day 2
  The plasma concentration level of brivaracetam 5 minutes postdose on Day 2.
Brivaracetam (BRV) plasma concentration (at Day 5) | Day 5
  The plasma concentration level of brivaracetam 5 minutes postdose on Day 5.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (9):
- Japan (9):
  - Ep0118 116, Asaka
  - Ep0118 126, Bunkyō City
  - Ep0118 111, Hamamatsu
  - Ep0118 121, Itami
  - Ep0118 142, Kamakura
  - Ep0118 112, Kōshi
  - Ep0118 104, Shizuoka
  - Ep0118 138, Tsukuba
  - Ep0118 109, Yamagata

IPD SHARING:
Plan to Share IPD: No